CLINICAL TRIAL: NCT03576209
Title: Prospective Study on Effects of a Healthy Lifestyle Program on Health Outcomes in Older Adults.
Brief Title: Effects of a Healthy Lifestyle Program on Health Outcomes in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Julie Vanderlinden, Principal Investigator, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lekker Actief
Record Dates: First submitted 2018-04-29; First posted 2018-07-03 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Sleep; Quality of Life; Functional Ability; Well-being; Social Identity; Leadership; Social Support; Motivation
Keywords: Physical activity; sedentary behaviour; sleep; Quality of life; functional ability; well-being; Social identity and leadership; social support and motivation; Aged, older adults
MeSH Terms: conditions — Social Identification; Motor Activity

STUDY DESIGN:
Intervention Model Description: The described trial is a controlled before-and-after study. In this study, observations are made before and after the implementation of the intervention during 12 weeks, both in groups participating in the program (intervention group) and in groups who are not participating in the program (control groups).
  Observations are made in intervention and control groups. Participants of the intervention group are registered for participation in this health promotion program 'Lekker Actief' prior to the start of this trial. The control groups are composed of participants who are not participating in the program (not receiving any intervention) or the controls are waitlist controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): 12 week intervention
  Interventions: Behavioral: healthy lifestyle program
- Control Group (No Intervention): No walking program

INTERVENTIONS:
Behavioral: healthy lifestyle program — Participants (intervention group) are following a 12 week health promotion program. They will count daily steps by pedometers and participate in weekly organised walks (within socio-cultural organisation)
  Other Names: 12 week program 'Lekker Actief'
  Arms: Intervention Group

SUMMARY:
Medical condition or disease under investigation : Quantitative and qualitative aspects of sleep, quality of life, functional ability and well-being in older adults (>55years)

Purpose of clinical trial : To study the prospective effects of a healthy lifestyle program on quantitative and qualitative aspects of sleep, quality of life, functional ability and well-being in older adults.

Primary objective : Measure the effects of the intervention on quantitative and qualitative aspects of sleep

Secondary objective (s) : Measure the effects of the intervention on physical activity, quality of life, functional ability and well-being Social identity and leadership, social support and motivation

Trial Design : Intervention study : controlled before-and-after study

Sample Size : total sample size : 1.000 participants

Summary of eligibility criteria : Older adults aged above 55years

Included in intervention group : adults who are participating in the healthy lifestyle promotion program 'Lekker Actief', organized by OKRA

Included in control group : waitlist controls or controls (adults, members of OKRA, not participating in the health promotion program 'Lekker Actief')

Maximum duration of treatment of a subject :

* Start of Health promotion program 'Lekker Actief' : September 2018
* Measurements with accelerometers will start prior to the health promotion program 'Lekker Actief' : July 2018
* End of Health promotion program 'Lekker Actief' : December 2019
* Duration of Health promotion program 'Lekker Actief': 12 weeks
* Maximal duration : July 2018-December 2019

DETAILED DESCRIPTION:
This trial will consist of 3 visits : Pretest and posttest.

* Pretest measurements (week 0)

  o Accelerometry : a subsample of participants form intervention and control groups (n=400) will be asked to wear an accelerometer (type GT3X) during 7 entire days prior to baseline measurements. (Timing : July 2018-July 2019)

  o Baseline measurements : during the start up moment of the program all participants from intervention and control groups will be asked : (Timing : July 2018-July 2019)
  * To fill out the self-reported questionnaire (survey) : the survey is composed of existing validated scales : IPAQ, PSQI, SF-12, WEMWBS, HAQ-DI. (references of validated scales are provided in the 'outcome measures' section)
  * To perform a walk test over 20 meters in order to determine the individual stride length
  * To perform a 6 minute walking test in order to self-report perceived exertion and physical fitness (by Borg Scale) and to determine the individual entry level of the program (entry levels vary between 1-12)
  * To wear the Pedometer (Omron® Walking Style one 2.0) on a daily basis and register the amount of daily steps in their personal registration forms
* Posttest measurements (week 12)

  * Accelerometry : a subsample of participants form intervention and control groups (n=400) will be asked to wear an accelerometer (type GT3X®) during 7 days prior to posttest measurements. (Timing : September 2018 - December 2019)
  * Posttest measurements : at the end of the program all participants will be asked :

(Timing : September 2018 - December 2019)

* To fill out the self-reported questionnaire (survey). In addition to the pretest questionnaire, the validated scales ILI, Mael and Ashford (1992) and BREQ-3 will be added and will be filled out only by participants of the intervention groups
* To perform a 6 minute walking test in order to self-report perceived exertion and physical fitness (by Borg Scale)
* To inform the investigators on the amount of daily steps (measured with pedometer type : Omron® Walking Style one 2.0) during the 12 week program o Focus groups : a subsample will be invited to take part in focus groups. During these focus groups, participants will be encouraged to discuss the program and possible effects in small groups (5 participants per group). A semi-structured interview guide will be used to guide the discussions.

ELIGIBILITY:
Inclusion Criteria:

-aged 55+ years

Exclusion Criteria:

-Participants who are physically unable to participate in weekly meetings (PAR-Q : Physical activity readiness scale) (Thomas et al., 1992)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in sleep | Pretest (week 0), posttest (week 12) and follow up (month 15)
  Change in quantity of sleep : measured in minutes and hours by accelerometry and self-reported questionnaires (PSQI : Pittsburgh Sleep Quality Index (PSQI)) Change in quality of sleep : measured by self-reported questionnaire (PSQI)

SECONDARY OUTCOMES:
Change in objectively perceived physical activity | Pretest (week 0), posttest (week 12) follow up (month 15)
  Quantity : measured in minutes and hours by accelerometry
Change in subjectively perceived physical activity | Pretest (week 0), posttest (week 12) follow up (month 15)
  Quantity : measured by self-reported questionnaires (IPAQ : International Physical Activity Questionnaire)
change in quality of life | Pretest (week 0), posttest (week 12) follow up (month 15)
  measured by self-reported questionnaire (SF-12 : Short Form Health Survey)
change in functional ability | Pretest (week 0), posttest (week 12) follow up (month 15)
  measured by self-reported questionnaire (HAQ-DI : Health Assessment Questionnaire)
change in wellbeing | Pretest (week 0), posttest (week 12) follow up (month 15)
  well-being : measured by self-reported questionnaire (WEMWBS : Warwick-Edinburgh Mental Well-being scale)
Social identity and leadership | Pretest (week 0), posttest (week 12)
  measured by self-reported questionnaire (ILI : Identity Leadership Inventory)
motivation | Pretest (week 0), posttest (week 12)
  measured by self-reported questionnaire (BREQ3 : Behavioural Regulation In Exercise Questionnaire)
Social support | Pretest (week 0), posttest (week 12)
  measured by self-reported questionnaire (De Bourdeaudhuij & Salis, 2002)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Vanderlinden, phds, Principal Investigator — KU Leuven
Locations (1):
- KULeuven, Leuven, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
When intervention is finished, publication in peer reviewed journals is planned
Supporting Information: Study Protocol
Time Frame: Study protocol will be published after start of the trial
Access Criteria: by Principal Investigator

REFERENCES:
- [Derived] Vanderlinden J, Biddle GJH, Boen F, van Uffelen JGZ. To be well or not to be well: compositional associations of physical activity, sedentary behaviour and sleep with mental well-being in Flemish adults aged 55+ years. J Act Sedentary Sleep Behav. 2023 May 1;2(1):9. doi: 10.1186/s44167-023-00019-3. PMID 40217356
- [Derived] Vanderlinden J, Boen F, Puyenbroeck SV, van Uffelen JGZ. The effects of a real-life lifestyle program on physical activity and objective and subjective sleep in adults aged 55+ years. BMC Public Health. 2022 Feb 19;22(1):353. doi: 10.1186/s12889-022-12780-2. PMID 35183133